CLINICAL TRIAL: NCT02728817
Title: Evaluation of the Radial Artery Deviation And Reimplantation Technique for Primary Hemodialysis Access Creation: a Multicenter Randomized Controlled Trial
Brief Title: Evaluation of the Radial Artery Deviation And Reimplantation Technique for Primary Hemodialysis Access Creation
Acronym: RADAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-API-02
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: End-stage Renal Disease
Keywords: Vascular access; Hemodialysis; Arteriovenous fistula; Stenosis; Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula; Constriction, Pathologic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arteriovenous fistula (AVF) (Active Comparator): Patient receiving a traditional arteriovenous fistula at the wrist (end-cephalic vein to side-radial artery)
  Interventions: Procedure: End-cephalic vein to side-radial artery fistula creation
- RADAR (Experimental): Patient receiving an arteriovenous fistula at the wrist using the Radial Artery Deviation And Reimplantation technique (end-radial artery to side-cephalic vein)
  Interventions: Procedure: RADAR fistula creation

INTERVENTIONS:
Procedure: End-cephalic vein to side-radial artery fistula creation — * Circumferential dissection of the cephalic vein (4-5cm long)
  * Longitudinal arteriotomy (~10mm)
  * End-vein to side-artery anastomosis using 7-0 polypropylene continuous suture
  Arms: arteriovenous fistula (AVF)
Procedure: RADAR fistula creation — * Dissection of the anterior-medial aspect of the cephalic vein (~15mm) without grasping or clamping the venous wall
  * Circumferential dissection of the radial artery pedicle (5cm long) and ligation of collaterals with surgical microclips
  * Ligation and section of the radial artery (distal)
  * Longitudinal venotomy (~10mm)
  * End-artery to side-vein anastomosis using 7-0 polypropylene continuous suture
  Arms: RADAR

SUMMARY:
The Radial Artery Deviation And Reimplantation (RADAR) technique is a new approach for the construction of hemodialysis arteriovenous fistula. In this technique, the radial artery pedicle is deviated towards the minimally dissected cephalic vein at the wrist. The aim of this study is to compare the safety and efficacy of this technique with the traditional end-cephalic to side-radial arteriovenous fistula, currently used as a first line vascular access in hemodialysis patients.

The hypothesis is that the minimal dissection concept used in the RADAR inhibits venous juxta-anastomotic neointimal hyperplasia and stenosis, and lead to higher rates of maturation and patency.

DETAILED DESCRIPTION:
In current nephrology and vascular surgery guidelines, end-cephalic to side-radial arteriovenous fistula is the gold standard for primary vascular access creation. However, these wrist AVFs are recognized to have the worst patency of any autogenous vascular accesses. Outcome improvement is therefore urgent in the field of vascular access, which concerns a growing incident population of patients with end-stage renal disease requiring hemodialysis.

Primary AVF failure, including failure to mature, occurs in ~35-40% in just the first year, generally due to juxta-anastomotic stenosis. Many AVF subsequently require additional interventions to mature successfully. The primary patency for these AVFs is poor with 55% at 12 months.

Juxta-anastomotic neointimal hyperplasia typically occurs in the swing segment, e.g. the proximal vein mobilized to form the end-to-side anastomosis. This surgically-mobilized segment coincides both with turbulent flow as well as with devascularization of the vasa vasorum. These processes have been associated with endothelial cell activation and a dysfunctional phenotype. Therefore investigators hypothesized that surgical techniques which minimize venous dissection may improve fistula maturation and access patency.

Accordingly, investigators developed the "Radial Artery Deviation And Reimplantation (RADAR) technique." Instead of using a traditional end-vein to side-artery anastomosis, RADAR uses an end-artery to side-vein anastomosis, additionally coupled with minimal vessel dissection. Investigators extend conventional "no touch" techniques and advocate avoidance of any venous dissection or manipulation. Investigators minimize arterial dissection as well, by dissecting the radial artery pedicle, not the artery itself.

The aim of this study is to compare the safety and efficacy of this novel technique with the traditional radial-cephalic fistula in the setting of a multicenter randomized controlled trial. Besides traditional endpoints such as patency and reintervention rates, hand blood perfusion will be assessed with objective measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred by the nephrologist for the creation of a primary vascular access
* Clinical examination of both upper limbs showing on the same limb:

  * A cephalic vein at the distal third of the forearm
  * Radial pulse
  * Ulnar pulse
  * Positive Allen test (patent palmar arches)
* Preoperative arterial and venous duplex ultrasound examination of both limbs showing on the same limb :

  * A patent cephalic vein, ≥2mm in diameter at the distal 1/3 of the forearm, free from stenosis, ≥15cm in length
  * A patent on dominant radial artery, ≥2mm in diameter at the distal 1/3 of the forearm, free from stenosis and major calcifications
  * A patent ulnar artery, free from stenosis and major calcifications
  * A positive Allen's test with assessment of the retrograde flow (patent palmar aches)
* Digital pressure >50mmHg when occlusive compression is made on the radial artery and digital/brachial ratio >0.5

Exclusion Criteria:

* patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate of the access | at 12 months

SECONDARY OUTCOMES:
Assisted primary patency rate of the access | 6 & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Serge DECLEMY, MD, Principal Investigator — Vascular surgery, Nice University Hospital
Locations (4):
- France (4):
  - Polyclinique Notre Dame, Draguignan
  - Aphm, Marseille
  - CHU de Nice - Service de chirurgie vasculaire, Nice
  - Polyclinique Les Fleurs, Ollioules

IPD SHARING:
Plan to Share IPD: No